CLINICAL TRIAL: NCT04109573
Title: Function Following Laser for Anal Intraepithelial Neoplasia (FLAN)
Acronym: FLAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R&DCL1403
Record Dates: First submitted 2016-04-21; First posted 2019-09-30 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Anus Cancer; Fecal Incontinence; Anal Intraepithelial Neoplasia; Post Operative Pain
Keywords: laser ablation; anal intraepithelial neoplasia; AIN; fecal incontinence; anal function
MeSH Terms: conditions — Anus Neoplasms; Fecal Incontinence; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anorectal function post anal laser (Experimental): Intervention:
  Device: laser
  Interventions: Procedure: high resolution anal manometry

INTERVENTIONS:
Procedure: high resolution anal manometry — functional studies before and after anal laser ablation
  Other Names: endoanal ultrasound; gastrointestinal physiology

SUMMARY:
High-grade squamous intraepithelial lesions (HSIL) and anal cancer are rising in incidence and at highest risk are HIV positive men who have sex with men (MSM). This pilot study assessing anal function and patient-reported outcomes before and after laser ablation of HSIL will add to the evidence that such a therapy is an acceptable and safe treatment to offer in a preventative setting.We will be recruting HIV positive and negative MSM.

DETAILED DESCRIPTION:
High resolution anoscopy with targeted laser ablation is one of the therapies currently employed to treat HSIL of the anus to prevent progression to anal cancer. The functional outcome of this procedure has not previously been formally assessed.

HIV and negative positive MSM in whom HSIL has been detected will form the study population, as HSIL is prevalent in these patients and intervention is felt to be indicated. Functional assessments will be carried out prior to initial treatment and then repeated six months after laser ablation therapy. The structure, function and sensitivity of the anal canal will be evaluated using endoanal ultrasound, high-resolution anal manometry and anal mucosal electrosensitivity measurements respectively. Patient-reported outcomes will be assessed using questionnaires and semi-structured interviews at baseline, 4 weeks and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

MSM >18 years of age if HIV positive, CD4 count of over 350; if less, been on highly active antiretroviral treatment for at least 3 months Histologically proven high-grade squamous anal intraepithelial neoplasia lesion (HSIL) Anal canal disease with or without perianal disease Written informed consent

Exclusion Criteria:

Previous laser or other ablative treatment for HSIL (previous topical treatment is not excluded) Any treatment for HSIL in the previous six months Previous or current diagnosis of anal cancer Concurrent or previous (if severe) perianal inflammatory bowel disease, complex fistula or other significant perianal condition requiring surgery including fissures, current fistula in ano and Grade III or IV haemorrhoids Perianal sepsis Perianal disease only without anal canal HSIL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Manometric indices | Six months
  Changes in pressure vailues - resting pressure and maximum squeeze pressure compared to patient's own pre treatment values

SECONDARY OUTCOMES:
Anal mucosal sensitivity | 6 months
  Changes in sensitivity as measured against patients own pre treatment perception
Endoanal ultrasound abnormalities | 6 months
  Changes in endoanal ultrasound abnormalities compared to pre-treatment findings
Physical and psychological well-being | 4 weeks 6 months
  Qualitative subjective physical and psychological well-being 4 weeks and 6 months after procedure of laser mucosal ablation of AIN
Patient reported outcomes | 6 months
  Patient reported outcomes, particularly with regard to sexual function and bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Tamzin Cuming, FRCS, Study Director — Homerton University Hospital NHS Trust
Locations (1):
- Homerton University Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No